CLINICAL TRIAL: NCT05134701
Title: Dapagliflozin Post-Marketing Surveillance in Heart Failure Patients and Chronic Kidney Disease Patients
Brief Title: Dapagliflozin Post Marketing Surveillance in HF and CKD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1699R00007
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure; Chronic Kidney Disease
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This is an observational, non-interventional, single-arm multicenter study. The objectives of this study are to assess safety and effectiveness of Forxiga in a real world setting in patients who are prescribed with the study drug according to the newly approved indications in the Republic of Korea

DETAILED DESCRIPTION:
As part of a post-approval commitment, the Ministry of Food and Drug Safety (MFDS) of the Republic of Korea (hereinafter "Korea") requests a study to characterize the safety in patients treated with dapagliflozin by physicians in normal clinical practice settings.

In principle, all patients treated with the product in accordance with the newly updated local prescribing information for HF and/or CKD are eligible for the enrolment in this study. Product prescription and patient enrollment will depend on physicians' medical decision as per routine clinical practice. Patient follow-up will be 12 weeks or about 24 weeks (for long-term surveillance) and patients will be recruited over a period of 4 years after the new HFrEF indication approval by the local health authorities. This is due to the requirements from the local health authorities.

The primary objective of this study is to assess the safety profile of the product in Korean adult patients with heart failure (HF) and/or chronic kidney disease (CKD) in a real world setting under the approved indication(s) in Korea.

The secondary objective of this study is to examine the effectiveness of the product in Korean patients with 1) HF and/or 2) CKD in a real world setting under the approved indication(s) in Korea.

The exploratory objective of this study is to identify patients' baseline characteristics that might be associated with the safety and effectiveness of the product when prescribed under the newly approved indication(s) in Korean patients with 1) HF and/or 2) CKD during the 12 weeks or about 24 weeks of follow-up duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years old and older
* Patients eligible for the product treatment (i.e. on-label treatment) according to the newly approved HF and/or CKD label in Korea
* Provision of signed and dated written informed consent by the patient or legally acceptable representative

Exclusion Criteria:

* Participation in any interventional trial during the treatment with the product.
* Any off-label indications that are not in accordance with the newly approved label in Korea.
* Any contraindications for the use of the product (as described in the local prescribing information).
* Prior use of product, as per local MFDS guidance.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: On active study drug treatment according to the approved local label.
Sampling Method: Non-Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Incidence (%) of adverse events (AEs), serious AEs (SAEs), adverse drug reactions (ADRs), serious ADRs (SADRs), unexpected AEs/ADRs, unexpected SAEs, SADRs | 12weeks or 24weeks

SECONDARY OUTCOMES:
No worsening in NYHA class from baseline | 12 weeks or 24 weeks
No worsening in UACR category from baseline | 12 weeks or 24 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Research Site, Busan
  - Research Site, Changwon
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Iksan
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suncheon
  - Research Site, Suwon
  - Research Site, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D169900007_Redacted_CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1699R00007&attachmentIdentifier=c920ca4a-a0db-478f-b09e-e416c7b8e6fe&fileName=D169900007_Redacted_CSR_Synopsis.pdf&versionIdentifier=